CLINICAL TRIAL: NCT04775719
Title: Pilot Sensor Randomized Controlled Trial: Setting Expectations to Increase Satisfactory Outcomes After Total Knee Replacement
Acronym: SensorRCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 10488
Record Dates: First submitted 2021-02-01; First posted 2021-03-01 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Patient Satisfaction
Keywords: Wearable Sensors; Machine Learning; Satisfaction; Expectations; Total Knee Arthroplasty
MeSH Terms: conditions — Patient Satisfaction; Personal Satisfaction

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: Members of the care team and investigator will be blinded from knowing which study arm the patient is in and what their predicted functional ability is, to ensure standard of care is not influenced in any way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Outcome Prediction Group (Other): Patient-Specific Prediction of Functional Outcome and Standard Pre-Operative Total Knee Arthroplasty Information
  Interventions: Other: Patient-Specific Prediction of Functional Outcome; Other: Standard Pre-Operative Total Knee Arthroplasty Information
- Standard Care Group (Other): Standard Pre-Operative Total Knee Arthroplasty Information
  Interventions: Other: Standard Pre-Operative Total Knee Arthroplasty Information

INTERVENTIONS:
Other: Patient-Specific Prediction of Functional Outcome — Information sheet that describes whether a patient is more likely to improve on or maintain their current preoperative function.
  Arms: Outcome Prediction Group
Other: Standard Pre-Operative Total Knee Arthroplasty Information — Standard of care information that is routinely provided at patient preadmission appointments.

SUMMARY:
More than 70,000 total knee replacement procedures are performed annually in Canada, representing a growth of 17% over the past 5 years, with further increases anticipated due to an aging population. While total knee replacement offers improved quality of life for patients and is cost effective for the healthcare system, 20% of patients routinely report dissatisfaction with the procedure. Patient dissatisfaction has been strongly linked to unmet expectations of outcomes after the surgery, especially with respect to physical activity. Counselling patients on appropriate expectations has been suggested as a means to improve satisfaction. Recently, our group has developed a tool to predict the functional ability of an individual patient after total knee replacement. This tool employs machine learning to classify patients as more likely to maintain or improve function, based on a functional test performed in clinic while wearing a sensor system around each knee. Implementing this tool in clinic pre-operatively could assist in setting appropriate expectations for each patient. Our primary objective is to compare patient satisfaction scores at one year after total knee replacement in patients who were informed of their specific expected functional outcome compared to patients who were not informed of their predicted functional outcome. We hypothesize that patients who are given an informed expectation will have higher satisfaction scores. This in turn may decrease health system costs associated with additional clinic visits from dissatisfied patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with osteoarthritis scheduled to undergo primary total knee arthroplasty

Exclusion Criteria:

* prior knee surgery
* inflammatory arthritis
* neuromuscular disorder that impairs gait
* scheduled for bilateral total knee arthroplasty
* Cannot read, write, or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-16 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Patient Satisfaction | Pre-operation, 3-months, and 1-year post-operation
  Patients will complete the Knee Society Score (KSS) questionnaire. The primary outcome of interest from the KSS is the satisfaction section. There are five questions related to satisfaction, each with five options ranging from very dissatisfied (0 points) to very satisfied (8 points).

SECONDARY OUTCOMES:
Cost Effectiveness | At 2-weeks, 6-weeks, 3-months, and 1-year post-operation
  Patient-reported cost diary

OTHER OUTCOMES:
Local Knee Inflammation | Pre-operation and 1-year post-operation (imaging). Intra-operative (tissue biopsies)
  Imaging and tissue biopsies to grade level of inflammation of the knee
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Pre-operation and 1-year post-operation
  Patient-reported questionnaire to assess pain, stiffness, and function.
Measure of Intermittent and Constant Osteoarthritis Pain (ICOAP) | Pre-operation and 1-year post-operation
  Patient-reported questionnaire to assess experience with constant and intermittent pain.
Patient Global Assessment (PGA) | Pre-operation and 1-year post-operation
  Patient-reported scale question to measure global disease activity on a range of 0 (doing very well) to 10 (doing very poorly)
Global Rating of Change Scale (GROC) | Pre-operation and 1-year post-operation
  Patient-reported questionnaire to assess self-perceived improvement.
EuroQuol 5D (EQ-5D) | Pre-operation and 1-year post-operation
  Patient-reported questionnaire to assess health-related quality of life and is used for economic analysis.
UCLA Activity Score | Pre-operation and 1-year post-operation
  Patient-reported questionnaire to assess activity from range of 1 (completely wholly inactive) to 10 (regularly participates in impact sports).

CONTACTS AND LOCATIONS:
Overall Officials: Brent Lanting, Principal Investigator — Lawson Health Science Centre
Locations (1):
- London Health Science Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No